CLINICAL TRIAL: NCT07051681
Title: Effect of Gestational Diabetes Mellitus on Serum Hormone Levels and Human Milk Composition
Brief Title: Gestational Diabetes and Human Milk Composition Study
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Collaborators: Zeynep Kamil Maternity and Pediatric Research and Training Hospital (Other)
Responsible Party: Principal Investigator, Sule Aktac, Assoc. Prof. Dr., Marmara University
Other Study IDs: BDB-MILK-TRIAL-2025
Record Dates: First submitted 2025-06-26; First posted 2025-07-04 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Gestational Diabetes Mellitus (GDM)
Keywords: GDM; human milk; hormone; nutrition therapy; postpartum period; adiponectin; chemerin; dermcidin; insulin; ghrelin; leptin
MeSH Terms: conditions — Diabetes, Gestational; Insulin Resistance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Human milk Blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- GDM: Pregnant women with GDM
  Interventions: Other: Individualized Medical Nutrition Therapy

INTERVENTIONS:
Other: Individualized Medical Nutrition Therapy — Pregnant women with GDM received individualized nutrition therapy during pregnancy. No intervention was applied to the control group.

SUMMARY:
This study aims to compare hormone levels and milk composition in women with and without gestational diabetes through postpartum human milk and blood samples.

DETAILED DESCRIPTION:
Pregnant women with GDM who received medical nutrition therapy and healthy controls were evaluated on postpartum days 14 and 30. Human milk and blood samples, as well as 3-day food consumption records, were collected. Levels of insulin, adiponectin, leptin, ghrelin, chemerin, and dermcidin in blood and milk were measured and compared with macronutrient contents of milk.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary pregnant women with singleton pregnancies
* No complications or chronic diseases.

Exclusion Criteria:

* With pregnant and post-partum complications or chronic diseases
* Mothers who feed their babies with formula

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Voluntary pregnant women attending Zeynep Kamil Women and Children's Hospital obstetrics clinic.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Serum hormone levels | Postpartum day 14 and 30
  Measurement of insulin, adiponectin, leptin, ghrelin, chemerin, and dermcidin levels using ELISA in maternal blood serum
Human milk hormone levels | Postpartum day 14 and 30
  Measurement of insulin, adiponectin, leptin, ghrelin, chemerin, and dermcidin levels using ELISA in human milk samples

SECONDARY OUTCOMES:
Human milk energy and macronutrient content | Postpartum day 14 and 30
  Analysis of energy, protein, fat, and lactose content in milk

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University, Maltepe, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results (text, tables, figures, and appendices) will be shared after de-identification. Data will be available beginning 6 months after publication, to researchers who provide a methodologically sound proposal.
Supporting Information: CSR